CLINICAL TRIAL: NCT03214497
Title: Prospective Randomised Trial of the Protector™ Versus the Supreme® Laryngeal Mask Airway
Brief Title: Protector™ Versus Supreme® Laryngeal Mask Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Schulthess_Anä_11
Record Dates: First submitted 2017-06-28; First posted 2017-07-11 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Anesthesia
Keywords: laryngeal mask; Supreme; Protector
MeSH Terms: interventions — Mouth Protectors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protector group (Active Comparator): All patients collocated randomly to the Protector Group Primary and secondary outcome Parameters are studied
  Interventions: Device: Protector
- Supreme group (Placebo Comparator): All patients collocated randomly to the Supreme Group, Primary and secondary outcome Parameters are studied
  Interventions: Device: Supreme

INTERVENTIONS:
Device: Protector — All patients which are assigned to the Protector are studied with this laryngeal mask
  Arms: Protector group
Device: Supreme — All patients which are assigned to the Supreme are studied with this laryngeal mask
  Arms: Supreme group

SUMMARY:
The goal of this study is to compare the oropharyngeal leak pressure of the Protector Laryngeal mask with the Supreme laryngeal mask. Other secondary parameters will be studied.

DETAILED DESCRIPTION:
The OLP as the primary outcome measurement will be evaluated after insertion of the LMA in each group. We hypothesize that there will be a difference of 4 cm H2O between the 2 masks, because of the different material and slightly different form of the masks. Secondary outcomes will be measured after insertion of the LMA as by protocol. Finally postoperative airway morbidity will be evaluated 3 hours after removal of the LMA.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75
* ASA 1-3
* Operation on limbs
* written informed consent

Exclusion Criteria:

* known difficult airway
* anatomical abnormalities on airway, Larynx, oesophagus, stomach
* not fastened
* high aspiration risk
* patients with contraindication of laryngeal mask
* BMI >35 kg/m2
* patients with disease which impairs accurate Investigation of patient
* cardiovascular risk factors
* COPD
* acute disease where anaesthesia is in doubt
* no written consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
OLP | 5 minutes
  oropharyngeal leak pressure

SECONDARY OUTCOMES:
insertion | 5 minutes
  insertion of LMA
time of insertion | 5 minutes
  time of Insertion of LMA
Brimacombe score | 5 minutes
  Brimacombe score
respiratory pressure | 5 minutes
  maximum respiratory pressure for adequate ventilation
suctioning catheter | 5 minutes
  number needed of insertion of suctioning catheter
suctioning fluids | 5 minutes
  ml suctioned from suctioning catheter
CO2 | 5 minutes
  endtidal CO2
blood staining | 5 minutes
  visible blood staining after removal of the laryngeal mask
airway morbidity | 3 hours
  assess sore throat, neck pain

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Moser, MD, MBA, Principal Investigator — Schulthess Klinik
Locations (1):
- Christian Keller, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes